CLINICAL TRIAL: NCT07114848
Title: Comparative Efficacy of Tamsulosin and Solifenacin in Managing Double J Stent-Related Symptoms: A Randomized Clinical Study Using the USSQ Tool.
Brief Title: Comparing Tamsulosin and Solifenacin for Relieving Double J Stent Symptoms: Using the USSQ.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Liaquat National Hospital & Medical College (Other)
Responsible Party: Principal Investigator, Fareha Khan, Urology Resident, Liaquat National Hospital & Medical College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0996-2024-LNH-ERC
Record Dates: First submitted 2025-07-17; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Ureteral Stent-Related Symptom; Alpha Blocker; Anticholinergics; Ureter Calculi
Keywords: Tamsulosin vs solifenacin in improving stent related symptoms; Double J stent; Tamsulosin; solifencin; ureteral stent-related symptoms; ussq; alpha-blocker; anticholinergic; RCT; quality of life
MeSH Terms: interventions — Tamsulosin; Solifenacin Succinate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tamsulosin (Active Comparator): Group A received tamsulosin starting within 24 hours after stent placement.
  Interventions: Drug: Tamsulosin
- Solifenacin (Active Comparator): Group B received solifenacin starting within 24 hours after stent placement.
  Interventions: Drug: solifenacin

INTERVENTIONS:
Drug: Tamsulosin — Tamsulosin 0.4 mg once daily for 14 days
  Other Names: Tamsolin
  Arms: Tamsulosin
Drug: solifenacin — Solifenacin 5 mg once daily for 14 day
  Other Names: solifen
  Arms: Solifenacin

SUMMARY:
This study evaluates the effects of two medications-tamsulosin and solifenacin-on symptoms associated with double J (DJ) ureteral stents. The research is conducted among patients undergoing unilateral DJ stent placement for ureteric calculi or post-ureteroscopic lithotripsy. Participants are randomly assigned to receive either tamsulosin or solifenacin, and symptom severity is assessed using the Ureteral Stent Symptom Questionnaire (USSQ).

DETAILED DESCRIPTION:
Ureteral stents are widely used in urological procedures but are frequently associated with stent-related symptoms such as urinary urgency, pain, and reduced quality of life. These symptoms are believed to arise from mechanical irritation and bladder overactivity. Alpha-blockers and antimuscarinic agents are commonly prescribed to alleviate these effects. This study is designed to compare the effects of tamsulosin, an alpha-1 adrenergic receptor antagonist, and solifenacin, a muscarinic M3 receptor antagonist, in reducing DJ stent-related symptoms.

The study is a single-center, randomized clinical trial conducted at the Department of Urology, Liaquat National Hospital, Karachi. Sixty adult patients who undergo unilateral DJ stent placement for ureteric stones or after ureteroscopic lithotripsy are randomized into two equal groups. Group A receives tamsulosin 0.4 mg daily, and Group B receives solifenacin 5 mg daily. Symptom evaluation is performed on day 14 post-procedure using a culturally adapted version of the Ureteral Stent Symptom Questionnaire (USSQ), which assesses domains such as urinary symptoms, pain, general health, work performance, and sexual health.

The findings from this study aim to inform treatment decisions for managing stent-related symptoms in similar clinical populations.

ELIGIBILITY:
Inclusion Criteria:

* Age 20 to 50 years
* Undergoing unilateral DJ stenting for:
* Ureteric calculi
* Post-ureteroscopic lithotripsy

Exclusion Criteria:

* Bilateral stents
* History of LUTS or recurrent UTI
* Urological malignancy or bladder surgery
* Known hypersensitivity to alpha-blockers or anticholinergics
* Uncontrolled hypertension, cardiovascular instability
* Chronic liver or kidney disease
* Stent complications (migration, encrustation, infection)

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2024-06-13 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-03-30 (Actual)

PRIMARY OUTCOMES:
Change in total USSQ score | 14days post stent placement
  Total score on the Ureteral Stent Symptom Questionnaire (USSQ), assessing pain, urinary symptoms, general health, work performance, and sexual health.

SECONDARY OUTCOMES:
Urinary index score | 14days
Pain index score | 14days
General Health Index score | 14days
Work Performance Index Score | 14days
Sexual Function Index Score | 14days

CONTACTS AND LOCATIONS:
Locations (1):
- Liaquat National Hospital, Karachi, Pakistan, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-06-12): https://cdn.clinicaltrials.gov/large-docs/48/NCT07114848/Prot_SAP_000.pdf
  • Informed Consent Form (2024-06-12): https://cdn.clinicaltrials.gov/large-docs/48/NCT07114848/ICF_001.pdf